CLINICAL TRIAL: NCT04736082
Title: Safety and Suitability of an Infant Formula Manufactured From Extensively Hydrolysed Protein in Healthy Term Infants
Brief Title: Safety of an Infant Formula With Hydrolysed Protein in Term Infants
Acronym: HASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HiPP GmbH & Co. Vertrieb KG (Industry)
Collaborators: Waldkrankenhaus Protestant Hospital, Spandau (Other); Biofortis, Merieux NutriSciences (Industry); HungaroTrial (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 508917-2
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Growth
Keywords: Safety; Growth; Weight Gain; Infant Formula; Infants
MeSH Terms: conditions — Weight Gain | interventions — Protein Hydrolysates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group: Infant Formula with hydrolyzed protein (Experimental): Infants will receive the following infant formula: Infant formula manufactured from extensively hydrolyzed proteins and containing pre- and probiotics.
  Interventions: Other: Intervention Group: Infant Formula with hydrolyzed protein
- Control Group: Infant Formula with intact protein (Active Comparator): Infants will receive the following infant formula: Infant formula manufactured from intact proteins and containing pre- and probiotics.
  Interventions: Other: Control Group: Infant Formula with intact protein
- Breast Fed Group (No Intervention): Exclusively breast milk

INTERVENTIONS:
Other: Intervention Group: Infant Formula with hydrolyzed protein — Infants will receive infant formula during the first 120 days of life with optional follow up until 180 days of life (intervention formula manufactured from extensively hydrolysed whey protein).
  Arms: Intervention Group: Infant Formula with hydrolyzed protein
Other: Control Group: Infant Formula with intact protein — Infants will receive infant formula during the first 120 days of life with optional follow up until 180 days of life (control formula manufactured from intact cow's milk protein).
  Arms: Control Group: Infant Formula with intact protein

SUMMARY:
A multi-centre, randomised, double-blind, parallel-group, controlled, prospective, non-inferiority intervention clinical trial is performed to assess the safety and suitability of an infant formula manufactured from extensively hydrolysed protein by showing normal growth of healthy term infants during the first 120 days of life with an optional follow up until 180 days of life.

DETAILED DESCRIPTION:
Since many years the use of infant formulae manufactured from hydrolysed proteins are recommended for infants at risk for developing allergies if they cannot be exclusively breast-fed. Although the use of such formulae manufactured from hydrolysed protein is legally authorized according to the respective legal framework since many years (currently: Directive 2006/141/EC), the safety of each hydrolysed protein has to be substantiated by additional clinical data according to new legal requirements (Del. Regulation (EU) 2016/127). This study is intended to generate clinical safety data: demonstrating adequate growth of infants fed a formula manufactured from hydrolysed protein in comparison to infants fed a formula manufactured from intact protein. As formula manufactured from hydrolyzed proteins is known to have beneficial effects on gastrointestinal comfort, it is also fed to infants not at risk for developing allergies. Therefore, this study additionally investigates the impact of hydrolysed protein on gastrointestinal tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female term infants until 25 days of age from singleton pregnancies
* Gestational age ≥37+0 weeks until 41+6 weeks
* Birth weight between ≥3rd and ≤97th percentile per gestational age
* Infants whose parent(s) / legally authorized representative(s) have reached the legal age of consent
* Infants whose parent(s) / legally authorized representative(s) are capable of and willing to comply with the protocol and have signed the informed consent form in accordance with legal requirements
* Infant formula group

  * Infants of mothers, who could not breastfeed their healthy newborn babies for reasons not related to this study, or who decided despite the advice on the benefits of breastfeeding to start exclusive formula-feeding within the first 25 days of age of their infant.
  * Parent(s) / legally authorized representative(s) confirm their intention to feed their infant the investigational product as the only source of nutrition from 26 days of age onward through the duration of the main study (until 120 days of age), and agree that no other infant formula, drinks (water, tea, juice,…) or complementary foods will be introduced until the infant reaches the age of 120 days.
* Breastfeeding reference group

  * Infants of mothers, who decided to exclusively breastfeed their infant until at least 120 days of age
  * Parent(s) / legally authorized representative(s) confirm their intention to breastfeed their infant as the only source of nutrition, from 26 days of age onward throughout the duration of the main study (until 120 days of age), and agree that no other infant formula, liquids (water, tea, juice,…) or complementary foods will be introduced until the infant reaches the age of 120 days.

Exclusion Criteria:

* Infants whose biological parents or full siblings have a history of doctor's diagnosed atopic diseases (atopic dermatitis, hay fever, allergic asthma or rhinitis) and have been in medical treatment prior to or at enrolment visit
* Intensive care prior to or at enrolment visit
* Severe acquired or congenital illness, or chromosomal anomalies (if known) in infants that are expected to interfere with normal feed or growth
* Hypo- or hypertrophy <3rd or >97th percentile of birth weight per gestational age
* Infants under (ongoing) antibiotic treatment before or at enrolment visit longer than three days (72 hours)
* Infants requiring infant formula intake other than those specified in the protocol
* Feeding difficulties or infant formula intolerance
* Disease of parents that may have an impact on study conduct or that may have an influence on infant growth and feeding behaviour based on the investigator's opinion
* Recreational drug or alcohol intake by the mother during the last two trimesters of pregnancy
* Infants born to mothers with medical conditions which have an effect on the infants' gastrointestinal tract/ability to be fed and/or growth (e.g. insulin dependent diabetes mellitus)
* Participation in another clinical intervention study

Ages: 0 Days to 25 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Infant daily weight gain (in g/day) between 30 days and 120 days of age | 90 days duration

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jochum, PD Dr. med., Principal Investigator — Evangelisches Waldkrankenhaus Spandau, Berlin, Germany
Locations (1):
- Evangelisches Waldkrankenhaus Spandau, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided